CLINICAL TRIAL: NCT06818942
Title: Nomogram for Predicting Difficult Laparoscopic Appendectomy
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Zhan, Principal Investigator, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-094(K)
Record Dates: First submitted 2025-01-26; First posted 2025-02-11 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Emergencies
Keywords: Laparoscopic appendectomy; Surgical difficulty; Training program
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult laparoscopic appendectomy: (1) operative time more than 75% of the overall study cases (2) severe intraoperative vascular or uncontrolled bleeding (3) conversion to open approach
  Interventions: Other: Observations on preoperative and intraoperative factors influencing the difficulty of surgery
- Non-difficult laparoscopic appendectomy: the remaining of the entire study cases excluding the difficult cases
  Interventions: Other: Observations on preoperative and intraoperative factors influencing the difficulty of surgery

INTERVENTIONS:
Other: Observations on preoperative and intraoperative factors influencing the difficulty of surgery — Age, body mass index, gender, inflammatory indicators, previous history of abdominal surgery, underlying disease

SUMMARY:
No prior studies have stratified the difficulty of laparoscopic appendectomy (LA). The investigators aimed to investigate preoperative factors as indicators of difficult LAs based on the experience of surgical trainees and to develop a predictive model accordingly.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of surgical emergencies and laparoscopic appendectomy (LA) is usually attempted by surgical trainees. This study aim to explore the preoperative and intraoperative factors affecting the degree of surgical difficulty and to establish a model for validation, so that it can be subsequently replicated in training programs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute appendicitis
* Participants who underwent laparoscopic appendectomy

Exclusion Criteria:

* Participants refused or could not tolerate laparoscopic appendectomy
* Incomplete preoperative examination or missed information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed acute appendicitis, were willing to and suitable to undergo laparoscopic appendectomy (LA). Patients were well informed about the surgical procedure and were aware of the potential benefits and risks. Patient consented for us to use perioperative data.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative time | During surgery
  operative time was defined as the duration from incision to closure, and was collected from anesthesia record sheet
Number of participants with postoperative complications | through study completion, an average of 1 year
  Postoperative bleeding, surgical site infection and other complications
Hospitalization | 1 day of discharge
  days of hospitalization
Degree of pain | approximately 4 hours after surgery and on postoperative day 1
  pain intensity was assessed using a standard visual analogue score, with a score of 0 to 10 corresponding to no pain to the most severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data are available on request due to privacy or other restrictions. The data that support the findings of this study are available on request from Ling Zhan. The data are not publicly available due to them containing information that could compromise research participant privacy.